CLINICAL TRIAL: NCT03409003
Title: Orphan Europe Carbaglu® Surveillance Protocol
Status: Recruiting | Type: Observational
Sponsor: Nicholas Ah Mew (Other)
Collaborators: Boston Children's Hospital (Other); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor-Investigator, Nicholas Ah Mew, Principal Investigator, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Other Study IDs: UCDC5111
Record Dates: First submitted 2016-11-18; First posted 2018-01-24 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: N-acetylglutamate Synthase (NAGS) Deficiency
Keywords: urea cycle disorder
MeSH Terms: conditions — Urea Cycle Disorders, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to conduct post-marketing surveillance of carglumic acid (Carbaglu) to obtain long-term clinical safety information. Carglumic acid was approved by the United States Food and Drug Administration (FDA) for treatment of acute hyperammonemia due to N-acetylglutamate synthase (NAGS) deficiency. Much of the FDA-required data is already collected through the Longitudinal Study of Urea Cycle Disorders (RDCRN Protocol #5101). This study will collect additional data on adverse events (interim events), adverse reactions, pregnancy, and fetal outcomes.

DETAILED DESCRIPTION:
Among the urea cycle disorders, N-acetylglutamate synthase (NAGS) deficiency is the rarest type. In 2010, carglumic acid (Carabglu) was approved by the United States Food and Drug Administration (FDA) "as an adjunctive therapy for the treatment of acute hyperammonemia due to the deficiency of the hepatic enzyme NAGS, and as maintenance therapy for chronic hyperammonemia due to NAGS deficiency." As post-marketing requirements, the US FDA requests that Orphan Europe (OE) conduct:

1604-2: A registry of patients, with NAGS deficiency being treated with carglumic acid to obtain long-term clinical safety information. Data will include patient demographics, details of treatment with carglumic acid, other therapies for hyperammonemia, dietary protein management, clinical status, neurocognitive and psychomotor status, growth and development status, and adverse events. Information from this registry is submitted to the FDA annually (in annual reports) with a final report submitted at 15 years post-approval.

1604-3: A study of the effects of carglumic acid on pregnancy and fetal outcomes. This study can be performed as a sub-study within the registry for all patients with NAGS deficiency. Information on pregnancy and fetal outcomes should be submitted annually (in annual reports) with a final report submission at 15 years post-approval.

This patient registry or surveillance protocol will be facilitated by collaboration with the existing National Institutes of Health (NIH) sponsored Urea Cycle Disorders Consortium (UCDC) Longitudinal Study of Urea Cycle Disorders (RDCRN Protocol #5101) (including NAGS deficiency) in the United States. The Longitudinal Study is sponsored by the NIH and other philanthropic sources. It is an academically governed network with the objective to conduct a longitudinal multidisciplinary investigation of the natural history, morbidity and mortality in people with UCD. It therefore aims to collect data on all patients with NAGS deficiency in the US. Measures in the Longitudinal Study are compatible with a Carbaglu post-marketing study including: developmental outcome, medical history, interval medical history, adverse events (interim events), pregnancy history, physical exam, vital signs, laboratory evaluation, dietary history, and medication records. Additional data on drug related adverse events and pregnancy outcomes will is collected for OE for FDA reporting.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of NAGS deficiency or suspicion of NAGS deficiency
* Carbaglu intake for the treatment of NAGS
* Enrolled in the Longitudinal Study of Urea Cycle Disorders (RDCRN protocol #5101)

Exclusion Criteria:

* Cases of hyperammonemia caused by other urea cycle disorders
* Organic acidemia, lysinuric protein intolerance
* Mitochondrial disorders
* Congenital lactic acidemia,
* Fatty acid oxidation defects
* Primary liver disease will be excluded
* Individuals with extreme low birth weight (<1,500 grams) will be also excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Confirmed diagnosis of NAGS deficiency or suspicion of NAGS deficiency, taking Carbaglu for the treatment of NAGS, and enrolled in the Longitudinal Study of Urea Cycle Disorders (RDCRN protocol #5101)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-04; Primary Completion 2026-07 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Carbaglu related adverse events and adverse reactions | 15 years
  The primary outcome measure is to monitor adverse events and adverse reactions, which will be reported to the FDA to fulfill post-marketing surveillance requirements.

SECONDARY OUTCOMES:
Number of hyperammonemic events | 15 years
  The number of hyperammonemic events (ammonia > 100 umol/L) will be monitored in participants taking Carbaglu to ensure there are no significant adverse changes
IQ | 15 years
  IQ will be monitored in participants taking Carbaglu to ensure there are no significant adverse changes
Height | 15 years
  Height (cm) will be monitored in participants taking Carbaglu to ensure there are no significant adverse changes
Weight | 15 years
  Weight (kg) will be monitored in participants taking Carbaglu to ensure there are no significant adverse changes
Abnormal physical and neurological findings | 15 years
  Any abnormal physical and neurological findings reported will be investigated as potential adverse reactions/adverse events (see primary outcome measure). Investigators conducts a review of systems and indicates whether findings are normal, abnormal or not assessed. Each abnormal finding is coded using SNOMED codes.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Ah Mew, MD, Principal Investigator — Children's National Research Institute
Locations (3):
- United States (3):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Hospital Boston (UCDC New England Center), Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No
This is a post-marketing surveillance study being performed so that Orphan Europe (OE) can meet its post FDA approval reporting obligations. Data will be shared with OE who will then report to the FDA. There are no other plans to make this data available to other researchers.

REFERENCES:
- See also: 5111: Orphan Europe Carbaglu® Surveillance Protocol In Collaboration with the Longitudinal Study of Urea Cycle Disorders — https://www.rarediseasesnetwork.org/cms/ucdc/Get-Involved/Studies/5111